CLINICAL TRIAL: NCT04976231
Title: Immunophenotyping of Patients With MPS II Treated With Enzyme Replacement Therapy
Brief Title: MPS II Immunophenotyping
Status: Terminated | Type: Observational
Why Stopped: Low Enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108243
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: MPS II; Mucopolysaccharidosis II; Hunter Syndrome
Keywords: MPS II; Mucopolysaccharidosis II; Hunter Syndrome
MeSH Terms: conditions — Sudden Infant Death; Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment Naive: Subjects who are naïve to ERT and start treatment with idursulfase
- Treatment less than 3 years: Subjects who have received ERT for <3 years
- Treatment over 3 years: Subjects who have received ERT for 3 or more years

SUMMARY:
The purpose of this study is to investigate how participant's body's immune system responds to idursulfase, an enzyme replacement therapy (ERT) and find out which types of immune cells are involved in causing untoward responses to the ERT so that the investigators can relate the level of immune response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of Mucopolysaccharidosis type II (MPS II) or Hunter Syndrome based on enzyme activity and variant analysis.
* Subject who plan to receive or have received enzyme replacement therapy with idursulfase.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metabolic or Genetics Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Changes in the frequency of natural killer cells measured by flow cytometry | baseline, 1, 3, 6 months
Changes in level of circulation memory B cells measured by flow cytometry | baseline, 1, 3, 6 months
Changes in level of T follicular helper cells measured by flow cytometry | baseline, 1, 3, 6 months
Changes in distribution of helper T cells measured by flow cytometry | baseline, 1, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No